CLINICAL TRIAL: NCT03942978
Title: Reducing Structural Inequities in Heart Failure Management: An Approach to Improve the Quality of Heart Failure Care on the General Medicine Service: Longitudinal Equity Action Plan (LEAP)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Robert Boxer, MD, Principal Investigator, Brigham and Women's Hospital
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2019P000951
Record Dates: First submitted 2019-04-24; First posted 2019-05-08 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Intervention Model Description: Stepped Wedge Randomized Control Trial
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Longitudinal Equity Action Plan (LEAP) (Active Comparator): Heart failure patients admitted with a principal diagnosis of heart failure to general medicine service and admitted to a general medicine pod that is randomized to the intervention arm.
  Interventions: Other: Longitudinal Equity Action Plan
- Standard Care (No Intervention): Heart Failure patients admitted to a general medicine pod at our institution, which is not randomized to intervention arm. Patients will be treated for their heart failure as per standard of care while admitted to the hospital.

INTERVENTIONS:
Other: Longitudinal Equity Action Plan — Patients admitted to general medicine pod randomized to intervention will receive a Longitudinal Equity Action Plan (LEAP), which will include a program manager to ensure they are on appropriate medical therapy, that cardiology is consulted when appropriate, that patient is set up with appropriate follow-up appointment with cardiology, that transportation is set up for follow-up visits, and a post-discharge follow up call to remind patients of the appointment and identify any post-discharge issues. This is in addition to standard of care, and there will not be any drug or device interventions.
  Arms: Longitudinal Equity Action Plan (LEAP)

SUMMARY:
Recent institutional research has demonstrated that black and Latinx patients are significantly less likely to be admitted to cardiology and more likely to be admitted to general medicine for their inpatient heart failure (HF) care. Subsequent HF care on general medicine has been demonstrated to have worse outcomes including lower rates of follow-up with cardiology and higher readmission rates. Given this, this project is a institutional quality improvement initiative, with a stepped wedge design, with the aim to improve the quality of care for heart failure patients admitted to general medicine for their care, and improve discharge planning. General medicine services by hospital pods will be enrolled in a stepped wedge fashion to a Longitudinal Equity Action Plan (LEAP) which includes a standardized clinical management plan to ensure patients are on guideline-appropriate therapy, receive cardiology consultation if appropriate, are discharged when clinically appropriate, discharge planning and systematic follow up with cardiology, transportation support as needed for follow-up visits, post-discharge follow up to identify any post-discharge issues.

DETAILED DESCRIPTION:
I. Aims with respect to Health Equity in the Department of Medicine

AIM 1: To improve the quality of care for heart failure patients admitted to the General Medicine Service (GMS) Aim 1a. To increase adherence and uptake of guideline-directed medical therapy and appropriate post-discharge follow-up for patients with heart failure admitted to GMS Aim 1b. To decrease 7-day heart failure readmission rates for patients with heart failure admitted to GMS with a principal diagnosis of heart failure Aim 1c. To decrease 30-day heart failure readmission rates for patients with heart failure admitted to GMS with a principal diagnosis of heart failure

AIM 2: To improve post-discharge outpatient cardiology utilization for heart failure patients admitted to GMS Aim 2a. To increase rates of cardiology clinic follow-up within 14 days of discharge for patients admitted to GMS with a principal diagnosis of heart failure.

II. Significance & Innovation A recent retrospective analysis performed by the Brigham and Women's Hospital (BWH) Cardiovascular Inequities Subcommittee of the Department of Medicine Health Equity Committee of patients self-referred to the Emergency Department with a principal diagnosis of heart failure found that black and Latinx patients were significantly less likely to be admitted to the cardiology service despite adjustment for multiple medical and socioeconomic factors (adjusted odds ratio [AOR] 0.68, 95% CI 0.53-0.87, for black patients; AOR 0.52, 95% CI 0.34-0.82 for Latinx patients). Female gender (AOR 0.75, 95% CI 0.62-0.91) and age>75 (AOR 0.58, 95% CI 0.40-0.86) were also independently associated with lower rates of admission to the cardiology service.

Similar to large observation studies from both community and academic settings, further analysis by the committee revealed differential outcomes for patients receiving specialty cardiology care during admissions for heart failure with lower cardiology clinic follow-up (25% vs. 51%), and higher 7-day (15% vs 5%) and 30-day (24 vs 17%) readmission rates for heart failure patients admitted to GMS as compared to those admitted to the cardiology service.

Given this result, the investigators hypothesize that inequities in admission service triage of heart failure patients may drive intra-hospital racial disparities in quality of care, and subsequent clinical outcomes. This project's aim is to achieve more equitable care and reduce unacceptable inequities in heart failure management and outcomes. Acknowledging that cardiology beds are a limited resource, and that not every patient can be admitted to the cardiology service at the investigators' institution, this project seeks to improve the quality of care for heart failure patients admitted to GMS. The investigators believe that improving the quality of heart failure care on GMS, including more systematic cardiology follow up, will lower heart failure readmission rates for the investigators' institution. Furthermore, this project will likely also lead to more equitable admission patterns downstream and will increase future admission to the cardiology service when appropriate because of the significant influence of cardiology outpatient follow up on admission to the cardiology service (adjusted OR of 2.31 [1.87, 2.84]).

III. Implementation Plan

Study design:

The investigators will implement a stepped-wedge design to expand to GMS a model of standardized clinical assessment and management (SCAMP) for heart failure. To assess the effectiveness of the intervention, measurement of cardiology clinic follow-up within 14 days of discharge, as well as 7-day and 30-day readmission rates for patients with heart failure admitted to GMS will be performed at baseline, at each cross-over time point, and at the conclusion of the intervention.

Methods:

Previous studies have demonstrated that SCAMPs lead to improved outcomes and promote the delivery of high-quality, cost-effective care. The SCAMP proposed, which is currently utilized for patients admitted to the BWH cardiology service, incorporates components of the American Heart Association's "Get with the Guidelines," to ensure patients are on guideline-directed medical therapy. The SCAMP as implemented on GMS will be titled the Longitudinal Equity Action Plan (LEAP), and will include support services to ensure 1) heart failure medications are covered and affordable 2) systematic scheduling of follow-up cardiology clinic appointments, and 3) barriers to patient attendance of cardiology appointments are addressed (e.g. through provision of ride vouchers). A LEAP program assistant will be responsible for completing the web-based LEAP form for each heart failure patient admitted to GMS. These forms are designed to ensure that patients are on guideline-directed medical therapy, with discussions with the primary medical team to understand rationale if medical therapy is not optimized, and that patients are scheduled with cardiologist follow-up appointment within 14 days of discharge. The LEAP program assistant will provide heart failure education to each patient including importance of weighing themselves daily, fluid and salt restriction, and in collaboration with the primary team, a "rescue plan" will be made for each patient in case they gain weight before their follow-up appointment. The LEAP program assistant will also be responsible for calling each patient's pharmacy to ensure medications are covered by insurance prior to discharge. Transportation assistance will be provided for all heart failure patients admitted to GMS to use for transportation to cardiology follow-up appointments..

The investigators will implement the LEAP within the investigators' institution's eight GMS teams. These teams have similar team structures, including a hospitalist attending and medical residents or physician assistants. The implementation of the medicine service will be introduced over a one-year period following a stepped wedge design. At four sequential time points, two GMS teams (clusters) will be randomized to cross from the usual care period to the intervention period. The process will continue until all clusters have crossed over to be exposed to the intervention (the LEAP). The intervention implementation process will include intensive training of hospital attendings, medical residents, and physician assistants in utilization of the LEAP.

Analysis:

The primary outcome of interest measured will be rates of cardiology clinic follow-up within 14 days. Second outcomes will include cardiology clinic follow-up within 30 days of discharge, 7-day readmission rates, and 30- day readmission rates. Other outcomes will include rates of cardiology consultation and rates of transportation support. The main analysis of the stepped wedge design will be based on a logistic mixed-effects model which will contain a random intercept to account for between-cluster variability, a fixed effect parameter for time, and a group indicator variable for the treatment for each subject and time to capture treatment differences over time. Assuming there are 20 patients per cluster, four time-points with one baseline measurement, and eight clusters, the investigators will have 98% power to detect a change in proportion of patients with 14-day cardiology follow-up from 25% to 50%, with Type I error rate of 5%.

IV. Future Directions and Amplification of Impact The investigators believe that improving heart failure care on GMS will lead to more equitable care and outcomes for not only black and Latinx patients but for all patients admitted to GMS with heart failure. If implementation of the LEAP on GMS proves to be impactful in improving heart failure outcomes, this may lead to uptake of similar strategies to improve care for other common disease entities, as well as access to specialized outpatient care, which is of paramount importance given that racial differences in referral patterns to outpatient specialty care for black and Latinx patients has been demonstrated. Success of this project may promote similar approaches to be employed by other departments to promote more equitable care of all patients. Furthermore, the investigators believe that this project will provide a platform for health equity capacity building for DOM faculty, opportunities for scholarship, and shared learning on health equity methodology.

ELIGIBILITY:
Inclusion Criteria:

* All patients admitted to the general medicine service at our hospital with a principal diagnosis of heart failure

Exclusion Criteria:

* Patients less than 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2019-05-31 (Actual); Primary Completion 2020-05-31 (Actual); Study Completion 2020-08-31 (Actual)

PRIMARY OUTCOMES:
Cardiology post-discharge follow-up within 14 days | 14 days
  Rates of patients that complete post-discharge follow up appropriate with a cardiologist within 14 days of discharge

SECONDARY OUTCOMES:
Seven-day Heart Failure Readmission | 7 days
  Rate of 7-day HF readmissions
30-day Heart Failure Readmission | 30 days
  Rate of 30-day HF Readmissions
Cardiology post-discharge follow-up within 30 days | 30 days
  Rates of patients that complete post-discharge follow up appropriate with a cardiologist

OTHER OUTCOMES:
Cardiology Consultation | Within admission
  Rates of cardiology consultation
Transportation Support | Within 14 days of discharge
  Rates of post-discharge follow up visit Transportation Support

CONTACTS AND LOCATIONS:
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yancy CW, Jessup M, Bozkurt B, Butler J, Casey DE Jr, Drazner MH, Fonarow GC, Geraci SA, Horwich T, Januzzi JL, Johnson MR, Kasper EK, Levy WC, Masoudi FA, McBride PE, McMurray JJ, Mitchell JE, Peterson PN, Riegel B, Sam F, Stevenson LW, Tang WH, Tsai EJ, Wilkoff BL. 2013 ACCF/AHA guideline for the management of heart failure: executive summary: a report of the American College of Cardiology Foundation/American Heart Association Task Force on practice guidelines. Circulation. 2013 Oct 15;128(16):1810-52. doi: 10.1161/CIR.0b013e31829e8807. Epub 2013 Jun 5. No abstract available. PMID 23741057
- [Background] Masters J, Morton G, Anton I, Szymanski J, Greenwood E, Grogono J, Flett AS, Cleland JG, Cowburn PJ. Specialist intervention is associated with improved patient outcomes in patients with decompensated heart failure: evaluation of the impact of a multidisciplinary inpatient heart failure team. Open Heart. 2017 Mar 8;4(1):e000547. doi: 10.1136/openhrt-2016-000547. eCollection 2017. PMID 28409010
- [Background] Jong P, Gong Y, Liu PP, Austin PC, Lee DS, Tu JV. Care and outcomes of patients newly hospitalized for heart failure in the community treated by cardiologists compared with other specialists. Circulation. 2003 Jul 15;108(2):184-91. doi: 10.1161/01.CIR.0000080290.39027.48. Epub 2003 Jun 23. PMID 12821540
- [Background] Foody JM, Rathore SS, Wang Y, Herrin J, Masoudi FA, Havranek EP, Krumholz HM. Physician specialty and mortality among elderly patients hospitalized with heart failure. Am J Med. 2005 Oct;118(10):1120-5. doi: 10.1016/j.amjmed.2005.01.075. PMID 16194643
- [Background] Salata BM, Sterling MR, Beecy AN, Ullal AV, Jones EC, Horn EM, Goyal P. Discharge Processes and 30-Day Readmission Rates of Patients Hospitalized for Heart Failure on General Medicine and Cardiology Services. Am J Cardiol. 2018 May 1;121(9):1076-1080. doi: 10.1016/j.amjcard.2018.01.027. Epub 2018 Feb 7. PMID 29548676
- [Background] Uthamalingam S, Kandala J, Selvaraj V, Martin W, Daley M, Patvardhan E, Capodilupo R, Moore S, Januzzi JL Jr. Outcomes of patients with acute decompensated heart failure managed by cardiologists versus noncardiologists. Am J Cardiol. 2015 Feb 15;115(4):466-71. doi: 10.1016/j.amjcard.2014.11.034. Epub 2014 Dec 2. PMID 25637324
- [Background] Selim AM, Mazurek JA, Iqbal M, Wang D, Negassa A, Zolty R. Mortality and readmission rates in patients hospitalized for acute decompensated heart failure: a comparison between cardiology and general-medicine service outcomes in an underserved population. Clin Cardiol. 2015 Mar;38(3):131-8. doi: 10.1002/clc.22372. Epub 2015 Feb 18. PMID 25694226
- [Background] Farias M, Jenkins K, Lock J, Rathod R, Newburger J, Bates DW, Safran DG, Friedman K, Greenberg J. Standardized Clinical Assessment And Management Plans (SCAMPs) provide a better alternative to clinical practice guidelines. Health Aff (Millwood). 2013 May;32(5):911-20. doi: 10.1377/hlthaff.2012.0667. PMID 23650325
- [Background] Hussey MA, Hughes JP. Design and analysis of stepped wedge cluster randomized trials. Contemp Clin Trials. 2007 Feb;28(2):182-91. doi: 10.1016/j.cct.2006.05.007. Epub 2006 Jul 7. PMID 16829207
- [Background] Cook NL, Ayanian JZ, Orav EJ, Hicks LS. Differences in specialist consultations for cardiovascular disease by race, ethnicity, gender, insurance status, and site of primary care. Circulation. 2009 May 12;119(18):2463-70. doi: 10.1161/CIRCULATIONAHA.108.825133. Epub 2009 Apr 27. PMID 19398667
- [Result] Caitlin S. Drescher, Kathryn A. Britton, Lynne W. Stevenson, Akshay S. Desai. Clinical Outcomes during Generalist Vs. Subspecialty Care of Inpatients with Heart Failure and Preserved Ejection Fraction. Journal of Cardiac Failure. 2017; 23(8):S23.